CLINICAL TRIAL: NCT04487561
Title: Hemopatch Versus Axillary Drainage After Axillary Lymphadenectomy: Randomized, Controlled, Multicenter Clinical Study
Brief Title: Hemopatch Versus Axillary Drainage After Axillary Lymphadenectomy
Acronym: REDHEMOPACH
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fundación para la Investigación del Hospital Clínico de Valencia (Other)
Responsible Party: Principal Investigator, Elvira Buch, Principal Investigator, Fundación para la Investigación del Hospital Clínico de Valencia
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: REDHEMOPACH
Record Dates: First submitted 2020-07-07; First posted 2020-07-27 (Actual); Last update posted 2023-02-17 (Actual); Status verified 2023-02

CONDITIONS: Breast Cancer; Breast-conserving Surgery; Axillary Lymph Node Dissection
Keywords: aspirative drainage; hemopatch; seroma; breast cancer
MeSH Terms: conditions — Breast Neoplasms; Seroma

STUDY DESIGN:
Intervention Model Description: Prospective multicentric randomized controlled clinical trial
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- aspirative drainage (Other): Drainage is the usual treatment after axillary lymphadenectoma for breast cancer
  Interventions: Procedure: Aspirative drainage
- Hemopatch (Active Comparator): The hemopatch group will be the group without drainage and with a product patch
  Interventions: Device: hemopatch

INTERVENTIONS:
Device: hemopatch — The patient will be randomized after performing the lymphadenectomy, according to a table of random numbers performed in excel kuytools, then a compression bandage will be performed on all the patients and it will be controlled 24 hours postoperatively, the subsequent control will be weekly until the drain is removed. and / or the disappearance of the seroma
  Arms: Hemopatch
Procedure: Aspirative drainage — The patient will be randomized after performing the lymphadenectomy, according to a table of random numbers performed in excel kuytools, then a compression bandage will be performed on all the patients and it will be controlled 24 hours postoperatively, the subsequent control will be weekly until the drain is removed. and / or the disappearance of the seroma
  Arms: aspirative drainage

SUMMARY:
Aspirative drainage continues to be the "gold standard" for the management of this post-surgical complication, even though it can lead to complications such as obstruction of the drainage, peritubal leakage of the seroma, etc. This may result in pain and reduction in mobility of the affected arm.

Based on our positive clinical outcomes and the fact that there is not any published data available in the literature regarding this use of the patch, the investigators propose a multicentric, randomized controlled clinical trial, with the objective of comparing the Hemopatch® with the usual technique used (aspirative drainage) in terms of efficacy and safety.

Hypothesis: Placing a Hemopatch ® instead of an aspirative drainage in women after undergoing axillary lymph node dissection during breast cancer surgery may reduce the appearance of seroma and consequently the need for a puncture, as well as the complications related to aspirative drainage.

DETAILED DESCRIPTION:
1. Introduction:

   In the surgical management of breast cancer, a conservative approach is the "gold standard" for the mammary region. For the axillary region, however, this depends on the results of the sentinel lymph node biopsy (SLNB) with axillary lymph node dissection (ALND) continuing to be an indispensable procedure when the disease reaches this level.

   The complications that arise from this procedure can be divided in two groups: 1) early: seromas and nerve lesions and 2) late: lymphedema, functional disorders in shoulder movement and post-mastectomy pain syndrome.

   Seromas are the most frequent complications after an ALND. In themselves, they do not carry a high risk of morbidity. However, they delay healing of the surgical wound, increasing the risk of infection and number of ambulatory visits and furthermore, resulting in a deferral in the start of adjuvant therapies such as radio and chemotherapy.

   Aspirative drainage continues to be the "gold standard" for the management of this post-surgical complication, even though it can lead to complications such as obstruction of the drainage, peritubal leakage of the seroma, etc. This may result in pain and reduction in mobility of the affected arm.

   Hemopatch® is a hemosthatic sealer made from reabsorbable collagen. It comes in the from of patch, with CE marking that is already being used in the clinical setting in Spain and the rest of Europe.

   Taking into account the factors that reduce seroma formation after ALND and the characteristics of the patch, its application after surgery could be useful in preventing seroma formation. More specifically, the patch has proven to act as a
   * Hemosthatic, improving the first phase of inflammation
   * Adhesive, reducing the dead space left after ALND
   * Sealer, decreasing the exudate
2. Rationale Based on this premise and in the context of a clinical protocol after the introduction of the patch in daily clinical practice, it was used on 28 patients that underwent ALND, obtaining favourable clinical results. This is a multicentric, randomized controlled clinical trial, with the objective of comparing the Hemopatch® with the usual technique used (aspirative drainage) in terms of efficacy and safety.
3. Hypothesis Placing a Hemopatch ® instead of an aspirative drainage in women after undergoing ALND during breast cancer surgery may reduce the appearance of seroma and consequently the need for a puncture, as well as the complications related to aspirative drainage.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of breast cancer,
* scheduled for surgical treatment including conservative surgery and ALND.
* Signed informed consent for ALND.

Exclusion Criteria:

* Selective sentinel node biopsy negative.
* Subsidiary mastectomy patients.
* Denial of informed consent for axillary lymphadenectomy.

Ages: 18 Years to 99 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 228 (Actual)
Dates: Start 2020-03-01 (Actual); Primary Completion 2023-02-14 (Actual); Study Completion 2023-02-14 (Actual)

PRIMARY OUTCOMES:
To develop seroma after surgery | Percentage, through study completion, an average of 2 months
  Percentage of patients that receive Hemopatch® that develop seroma after surgery and percentage of patients that receive that develop seroma after extraction of the aspirative drainage.
total volumen of the seroma | from 24 hours until there is no seroma, assessed up to 2 months
  The initial control will be performed 24 hours after the intervention, maintaining AD if the volume is greater than 30ml. All patients will be seen 7 days after surgery. The follow-up time will be weekly until there is no seroma, measuring the volume of the seroma extracted by puncture,
Seroma punctures | through study completion, an average of 2 months
  the total number of punctures needed
complications | from 24 hours until there is no complications, assessed up to 2 months
  Other complications collected throughout the study include: bruising (yes / no), pain (yes / no), problems with aspiration drainage (yes / no)

SECONDARY OUTCOMES:
quality of life in patients | 1 week after surgery with Eortc QLQ-BR23
  Compare the quality of life in patients after receiving either of these procedures using the Eortc QLQ-BR23 survey
the costs | through study completion, an average of 1 year
  Compare the costs of both procedures by quantifying the costs of materials and consult time used in both procedures
body mass index | weight (kg) / height (m2). In the first consultation
  body mass index

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Clínico Universitario de Valencia, Valencia, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lewis KM, Ikeme S, Olubunmi T, Kuntze CE. Clinical effectiveness and versatility of a sealing hemostatic patch (HEMOPATCH) in multiple surgical specialties. Expert Rev Med Devices. 2018 May;15(5):367-376. doi: 10.1080/17434440.2018.1464909. Epub 2018 Apr 26. PMID 29658322
- [Background] Droeser RA, Frey DM, Oertli D, Kopelman D, Baas-Vrancken Peeters MJ, Giuliano AE, Dalberg K, Kallam R, Nordmann A. Volume-controlled vs no/short-term drainage after axillary lymph node dissection in breast cancer surgery: a meta-analysis. Breast. 2009 Apr;18(2):109-14. doi: 10.1016/j.breast.2009.02.003. Epub 2009 Mar 16. PMID 19289285
- [Background] Aitken DR, Minton JP. Complications associated with mastectomy. Surg Clin North Am. 1983 Dec;63(6):1331-52. doi: 10.1016/s0039-6109(16)43192-0. No abstract available. PMID 6359504
- [Background] Kottayasamy Seenivasagam R, Gupta V, Singh G. Prevention of seroma formation after axillary dissection--a comparative randomized clinical trial of three methods. Breast J. 2013 Sep-Oct;19(5):478-84. doi: 10.1111/tbj.12164. Epub 2013 Jul 19. PMID 23865902
- [Background] Weber WP, Tausch C, Hayoz S, Fehr MK, Ribi K, Hawle H, Lupatsch JE, Matter-Walstra K, Chiesa F, Dedes KJ, Berclaz G, Lelievre L, Hess T, Guth U, Pioch V, Sarlos D, Leo C, Canonica C, Gabriel N, Zeindler J, Cassoly E, Andrieu C, Soysal SD, Ruhstaller T, Fehr PM, Knauer M; Swiss Group for Clinical Cancer Research (SAKK). Impact of a Surgical Sealing Patch on Lymphatic Drainage After Axillary Dissection for Breast Cancer: The SAKK 23/13 Multicenter Randomized Phase III Trial. Ann Surg Oncol. 2018 Sep;25(9):2632-2640. doi: 10.1245/s10434-018-6556-9. Epub 2018 Jun 8. PMID 29948418
- [Background] He XD, Guo ZH, Tian JH, Yang KH, Xie XD. Whether drainage should be used after surgery for breast cancer? A systematic review of randomized controlled trials. Med Oncol. 2011 Dec;28 Suppl 1:S22-30. doi: 10.1007/s12032-010-9673-2. Epub 2010 Sep 9. PMID 20827578
- [Background] Thomson DR, Sadideen H, Furniss D. Wound drainage after axillary dissection for carcinoma of the breast. Cochrane Database Syst Rev. 2013 Oct 20;2013(10):CD006823. doi: 10.1002/14651858.CD006823.pub2. PMID 24158902
- [Background] Petrek JA, Blackwood MM. Axillary dissection: current practice and technique. Curr Probl Surg. 1995 Apr;32(4):257-323. doi: 10.1016/s0011-3840(05)80015-2. No abstract available. PMID 7705102
- [Background] Kuroi K, Shimozuma K, Taguchi T, Imai H, Yamashiro H, Ohsumi S, Saito S. Pathophysiology of seroma in breast cancer. Breast Cancer. 2005;12(4):288-93. doi: 10.2325/jbcs.12.288. PMID 16286909
- [Background] Bonnema J, Ligtenstein DA, Wiggers T, van Geel AN. The composition of serous fluid after axillary dissection. Eur J Surg. 1999 Jan;165(1):9-13. doi: 10.1080/110241599750007441. PMID 10069628
- [Background] McCaul JA, Aslaam A, Spooner RJ, Louden I, Cavanagh T, Purushotham AD. Aetiology of seroma formation in patients undergoing surgery for breast cancer. Breast. 2000 Jun;9(3):144-8. doi: 10.1054/brst.1999.0126. PMID 14731838
- [Background] Lotze MT, Duncan MA, Gerber LH, Woltering EA, Rosenberg SA. Early versus delayed shoulder motion following axillary dissection: a randomized prospective study. Ann Surg. 1981 Mar;193(3):288-95. doi: 10.1097/00000658-198103000-00007. PMID 7011221
- [Background] Pinero-Madrona A, Castellanos-Escrig G, Abrisqueta-Carrion J, Canteras-Jordana M. Prospective randomized controlled study to assess the value of a hemostatic and sealing agent for preventing seroma after axillary lymphadenectomy. J Surg Oncol. 2016 Sep;114(4):423-7. doi: 10.1002/jso.24344. Epub 2016 Jun 23. PMID 27338717
- [Background] Conversano A, Mazouni C, Thomin A, Gaudin A, Fournier M, Rimareix F, Bonastre J. Use of Low-Thrombin Fibrin Sealant Glue After Axillary Lymphadenectomy for Breast Cancer to Reduce Hospital Length and Seroma. Clin Breast Cancer. 2017 Jul;17(4):293-297. doi: 10.1016/j.clbc.2016.12.013. Epub 2017 Jan 10. PMID 28161131
- [Background] Vasileiadou K, Kosmidis C, Anthimidis G, Miliaras S, Kostopoulos I, Fahantidis E. Cyanoacrylate Adhesive Reduces Seroma Production After Modified Radical Mastectomy or Quadrantectomy With Lymph Node Dissection-A Prospective Randomized Clinical Trial. Clin Breast Cancer. 2017 Dec;17(8):595-600. doi: 10.1016/j.clbc.2017.04.004. Epub 2017 Apr 13. PMID 28673765
- [Derived] Buch-Villa E, Castaner-Puga C, Delgado-Garcia S, Fuster-Diana C, Vidal-Herrador B, Ripoll-Orts F, Galeote-Quecedo T, Prat A, Andres-Matias M, Jimeno-Fraile J, Munoz-Sorsona E, Vento G, Gumbau-Puchol V, Adrianzen M, Lopez-Flor V, Ortega J. Clinical and cost outcomes of a polyethylene glycol (PEG)-coated patch versus drainage after axillary lymph node dissection in breast cancer: results from a multicentre randomized clinical trial. Br J Surg. 2023 Aug 11;110(9):1180-1188. doi: 10.1093/bjs/znad150. PMID 37311694
- See also: Survey of Eortc QLQ- BR23 — http://www.eortc.org
- See also: Pathophysiology of seroma in breast cancer. Breast Cancer [Internet]. 2005;12(4):288-93. — http://www.ncbi.nlm.nih.gov/pubmed/16286909